CLINICAL TRIAL: NCT01355510
Title: Electrical Baroreflex Stimulation - Sympathetic Activity
Brief Title: Effects of Electrical Baroreflex Stimulation on Sympathetic Activity, Renal Hemodynamics, and Insulin Sensitivity
Acronym: CVRX-ReSy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: DE-MHH-CVRX-ReSy-EK5753
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Electrical stimulation of carotid baroreceptors (baropacing) acutely decreases arterial pressure in patients with refractory hypertension. The reduction in blood pressure seems to be mediated through sympathetic inhibition with concomitant reduction in the activity of the renin-angiotensin system. Indeed, switching on and off the stimulation is accompanied by decreases and increases in central sympathetic vasoconstrictor outflow, respectively. Plasma renin concentration also decreases with acute electrical baroreflex stimulation.

In some patients chronic baropacing is associated with long-term blood pressure reduction.

However, there is sparse information as to the relative contribution of blood pressure regulating systems to account for the acute and chronic effects of baropacing. Sympathetic, renal, and vascular mechanisms are of special interest. Furthermore, technical aspects of electrical baroreflex stimulation may play a role, e.g. worsening of the electrical contact between the stimulating electrodes and the baroreceptor afferents.

This study is designed to answer the following primary questions:

1. Does chronic electrical stimulation of carotid baroreceptors inhibit sympathetic vasoconstrictor tone also in the long-term?
2. Does sympathetic vasoconstrictor tone increase on switching off chronic baropacing? Such an increase would confirm electrical integrity of the system and proper contact to the baroreceptor afferents.
3. Does acute electrical baroreflex stimulation decrease renal vascular resistance?
4. Does acute electrical baroreflex stimulation influence glucose delivery to skeletal muscle and change insulin sensitivity? The study follows an open-label observational design and it is planned to recruit up to 30 patients over 3 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment in the study:

* Adult patients having an implanted device for electrical baroreflex stimulation.
* Signed written informed consent.

Exclusion Criteria:

Subjects meeting all of the following criteria will be excluded from the study:

ReSy Study - Protocol version: December 20, 2010 8

* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Subject unlikely to comply with protocol, e. g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Pregnancy. Breast-feeding.
* History of hypersensitivity to inulin or paraaminohippurate or to drugs with a similar chemical structure have to be excluded from the constant-infusion procedure.
* History of drug or alcohol abuse.
* Blood donation of more than 500 mL during the previous 3 months (men) or 6 months (women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with implanted devices for electrical baroreflex stimulation are recruited according to inclusion and exclusion criteria until good quality recordings have been obtained in 20 patients during both stimulator settings (ON and OFF) in the corresponding study arm. After obtaining written informed consent patients will be investigated in the laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany